CLINICAL TRIAL: NCT05555459
Title: The Performance and Safety Evaluation of Bioabsorbable Headless Inion CompressOn Screws in Selected Fracture, Osteotomy and Artrodesis Surgeries of the Foot and Ankle
Brief Title: Performance and Safety Evaluation of Inion CompressOn Screw in Foot and Ankle Surgeries. PMCF Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inion Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CompressOn1-2022
Record Dates: First submitted 2022-09-08; First posted 2022-09-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Medial Malleolus Fracture; Lisfranc Injury; Lisfranc Fracture; Talus Fracture; Calcaneus Fracture; Navicular Fracture; Deformity, Foot; Ankle Fractures; Foot Fracture; Fractures, Bone; Fracture of Foot; Foot Deformities; Foot Injury; Feet Deformity Tarsus; Metatarsalgia; Hallux Rigidus; Hallux Valgus; Deformity of Toe; Deformity of Foot
Keywords: bioabsorbable screw; compression screw; headless screw; orthopaedic screw; bone fixation; bioabsorbable screw study; resorbable; biodegradable; bioabsorbable; fracture fixation with resorbable implants; inion; post-market follow-up study; orthopedic bone fixation; arthrodesis; osteotomy
MeSH Terms: conditions — Ankle Fractures; Foot Deformities; Fractures, Bone; Foot Injuries; Metatarsalgia; Hallux Rigidus; Hallux Valgus; Ankylosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A single group study including 125 adult patient participants. All patients undergo a bone fixation surgical operation in foot/ankle area. Indications are specified in the study description. All operations are performed in the one study center using Inion CompressOn screws.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CompressOn group (Experimental): 125 participant patients undergoing bone fixation surgical operation specified in the study description. All bone fixation surgeries are performed using Inion CompressOn screws.
  Interventions: Procedure: Operation

INTERVENTIONS:
Procedure: Operation — Bone fixation operation in foot or ankle area using bioabsorbable headless screw/s

SUMMARY:
The study in question is a post market clinical follow up (PMCF) study to evaluate the safety and performance of bioabsorbable headless compression screw Inion CompressOn in selected fracture, osteotomy and arthrodeses operations of the foot and ankle. The study recruits 125 adult patients who meet the acceptance criteria. The follow-up time for each study patient is 4 years. The study is a single center single group study which is conducted in Tampere University Hospital (TAYS) in Finland. The main focus of the study in terms of performance is to evaluate the bone healing/ossification of operated areas. The main focus of the study in terms of safety is to evaluate the occurrence of adverse events and required revision surgeries that are or might be related to the study device.

DETAILED DESCRIPTION:
The study in question is a post market clinical follow-up study to evaluate the safety and performance of bioabsorbable headless compression screw Inion CompressOn in selected fracture, osteotomy and arthrodeses operations of the foot and ankle. The main focus of the study in terms of performance is to evaluate the bone healing/ossification of operated areas. The main focus of the study in terms of safety is to evaluate the occurrence of adverse events and required revision surgeries that are or might be related to the study device.

The Inion CompressOn™ screws are cannulated headless compression screws made of degradable co-polymers composed of L-lactic acid and D-lactic acid. These polymers have a long history of safe medical use and they degrade in vivo by hydrolysis into alpha-hydroxy acids that are metabolised by the body. The screws retain their initial strength up to 12 weeks after implantation and gradually lose their strength thereafter. Bioabsorption takes place within two to four years. The Inion CompressOn™ products are intended for maintenance of alignment and fixation of bone fractures, comminuted fractures, osteotomies, arthrodeses or bone grafts (i.e., autografts or allografts) in the presence of appropriate additional immobilization (e.g., rigid fixation implants, cast or brace).

In the field of foot and ankle traumatology the surgical indications of this study include medial malleolar fractures, Lisfranc injuries, talus fractures, calcaneal fractures and navicular bone fractures. In the field of foot and ankle orthopaedics the surgical indications of the study include arthrodesis of the talonavicular joint, calcaneacuboideal joint, tarsometatarsal joint and first metatarsophalangeal (MTP1) joint, and osteotomies of the first metatarsal bone, second metatarsal bone (weil) and calcaneal bone.

The clinical data collection acquired from this study is a requirement of the EU Notified Body as part of the admitted CE mark certification, in cases when the device is initially approved based on the clinical data of an equivalent device. In this case, the equivalent device has been Inion FreedomScrew, which is made of the same material composition and has the same indications for use. Inion CompressOn Screw has new design features such as headless design, and threading which allows compression to the fracture line. Also new sizes are introduced.

The study recruits 125 adult patients who meet the acceptance criteria and have signed the informed consent. The follow-up time for each study patient is 4 years. Each patient has 6 follow-up time points related to the study. These time points consist of:

1. screening visit (-180-0 days before operation),
2. operation (day 0),
3. post-operative follow-up 1 (6 weeks after operation +/- 1 week),
4. post-operative follow-up 2 (3 months after operation +/- 2 weeks),
5. post-operative follow-up 3 (2 years after operation +/- 2 months)
6. post-operative follow-up 4 (4 years after operation +/- 4 months) The first 4 time points are within standard care, the last 2 time points (post-operative follow-up 3 and post-operative follow-up 4) are scheduled for study purposes only to be able to gain performance and safety data based on adequate follow-up time.

The study is a single center single group study which is conducted in Tampere University Hospital (TAYS) in Finland.

ELIGIBILITY:
Inclusion Criteria:

1. Read the patient information bulletin on the study and signed the patient consent form
2. Adult patient (over 18-year-old)
3. Suitable and in need for surgical lower limb operation listed in the indications of this study that requires fastening of bone structures with screws (or an alternative attachment method) in the ankle or foot area, according to a statement of the investigator surgeon
4. Ability to fill in questionnaires.
5. Willingness to comply with rehabilitation instructions.
6. Availability for follow-up visits.

Exclusion Criteria:

1. Active infection
2. Patient conditions including limited blood supply (e.g. patients with severe circulatory disorder of the lower limb
3. Patient conditions including insufficient quality or quantity of bone (diagnosed osteoporosis, conditions causing secondary osteoporosis e.g. diabetes, rheumatism, eating disorder)
4. Patient conditions where patient cooperation cannot be guaranteed (alcohol use, drug abuse etc.)
5. High-load bearing indications (e.g., diaphyseal fractures of long bones) unless used in conjunction with traditional rigid fixation
6. Patients with significant neuropathy
7. Pregnancy
8. Patients who refuse to participate
9. Lower limb tumor or metastasis
10. Complex Regional Pain Syndrome (CRPS) in operated foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Bone healing (ossification) of the fracture, osteotomy and arthrodesis lines | Change from operation to 4 years
  X-ray evaluation of bone healing (ossification) of the fracture, osteotomy and arthrodesis lines
Occurrence of adverse events (AEs) | During 4-year follow-up
  Assessment of occurrence of adverse events (AE), such as non-union of bone, fixation failure, mechanical irritation and tissue reactions related to implant bioabsorption
Occurrence of revision surgeries | During 4-year follow-up
  Assessment of occurrence of revision surgeries related to study device

SECONDARY OUTCOMES:
Subjective functionality of the operated foot or ankle (VAS foot and ankle) | Change from baseline to 4 years
  Evaluation of subjective pain of the operated foot or ankle during follow-up
Subjective functionality of the operated foot or ankle (EFAS) | Change from baseline to 4 years
  Evaluation of subjective functionality of the operated foot or ankle during follow-up
Wound and soft tissue healing | Change from operation to 3 months
  Assessment of post-operative complications (wound and soft tissue healing based on inspection and palpation)
Fixation strength | Change from operation to 4 years
  X-ray evaluation of the maintaining of fixation position
Bone formation in screw tunnel | Change from operation to 4 years
  X-ray evaluation of the level of bone formation in screw tunnel

CONTACTS AND LOCATIONS:
Overall Officials: Mäenpää, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No